CLINICAL TRIAL: NCT01275417
Title: Using Different Kinds of B-cun Scales to Mark Some Acupoints at Governor Vessel on the Head
Acronym: BCSM
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: Graduate Institute of Acupuncture Science, China Medical University (Other)
Responsible Party: China Medical University Graduate Institute of Acupuncture Science
Other Study IDs: DMRR99-IRB-152
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-01

CONDITIONS: to Research the Feasibility of the Proportional Bone(Skeletal) Measurement Method on the Head Region.
Keywords: Acupuncture

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- adult: 100 volunteers age ranged 18-80 years old
- children: 60 children under 10 years old.

SUMMARY:
We are expecting that there are remarkable differences location at BaiHui(GV20) or Houding(GV19)showing from same person in our study.

ELIGIBILITY:
Inclusion Criteria:

healthy volunteers

Exclusion Criteria:

1. craniectomy
2. Psychotic symptoms

Ages: 6 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sample: This experiment will recruit 100 volunteers age ranged 18-80 years old and 60 children under 10 years old.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)